CLINICAL TRIAL: NCT05835687
Title: Loc3CAR: Locoregional Delivery of B7-H3-specific Chimeric Antigen Receptor Autologous T Cells for Pediatric Patients With Primary CNS Tumors
Brief Title: Loc3CAR: Locoregional Delivery of B7-H3-CAR T Cells for Pediatric Patients With Primary CNS Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Loc3CAR; NCI-2023-02484 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2023-03-23; First posted 2023-04-28 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Central Nervous System Neoplasms; Atypical Teratoid/Rhabdoid Tumor; Diffuse Midline Glioma, H3 K27M-Mutant; Ependymoma; High Grade Glioma; Glioblastoma; Medulloblastoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Rhabdoid Tumor; Ependymoma; Glioma; Glioblastoma; Medulloblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (relapsed/refractory CNS tumors) (Experimental): Patients with B7-H3-positive relapsed/refractory non-brainstem primary CNS tumors.
  Interventions: Drug: B7-H3-CAR T cells
- Arm B (diffuse midline gliomas [DMG]) (Experimental): Patients with DMG.
  Interventions: Drug: B7-H3-CAR T cells

INTERVENTIONS:
Drug: B7-H3-CAR T cells — Autologous T cells transduced with a lentiviral vector expressing a B7-H3-CAR with a CD28z signaling domain and 41BB ligand (B7-H3-CAR T cells). Four (4) infusions of B7-H3-CAR T cells will be locoregionally administered via CNS reservoir catheter.

SUMMARY:
Loc3CAR is a Phase I clinical trial evaluating the use of autologous B7-H3-CAR T cells for participants ≤ 21 years old with primary CNS neoplasms. B7-H3-CAR T cells will be locoregionally administered via a CNS reservoir catheter. Study participants will be divided into two cohorts: cohort A with B7-H3-positive relapsed/refractory non-brainstem primary CNS tumors, and cohort B with diffuse midline gliomas (DMG). Participants will receive four (4) B7-H3-CAR T cell infusions over a 4 week period. The purpose of this study is to find the maximum (highest) dose of B7-H3-CAR T cells that are safe to give patients with primary brain tumors.

Primary objectives

* To determine the safety, maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) for the locoregional delivery of autologous B7-H3-CAR T cells in patients ≤ 21 years of age with recurrent/refractory B7-H3+ primary CNS tumors (Cohort A) or DMG (Cohort B).

Secondary objectives

* To assess the efficacy, defined as sustained objective response, a partial response (PR) or complete response (CR) observed anytime on active treatment with B7-H3-CAR T cells in patients with relapsed/refractory B7-H3+ primary CNS tumors (Cohort A) or DMG (Cohort B).
* To characterize and monitor neurologic toxicities in patients while on study (Cohort A and B).

DETAILED DESCRIPTION:
Treatment on this study includes four (4) B7-H3-CAR T cell infusions over a 4 week period. B7-H3-CAR T cells will be locoregionally administered via a CNS reservoir catheter without lymphodepleting chemotherapy. The study will evaluate the safety and maximum tolerated dose (MTD) of B7-H3-CAR T cells using a 3+3 study design and a 4 week evaluation period. Follow up will occur on this protocol for 1 year after the final B7-H3-CAR T cell infusion and then continue on an institutional long-term follow up protocol to complete 15 years post-infusion.

ELIGIBILITY:
Inclusion Criteria: Screening Eligibility

1. Age ≤ 21 years of age
2. Primary CNS tumor
3. For Cohort A, must have evidence of relapsed or refractory non-brainstem CNS tumor
4. For Cohort B, must meet one of the following criteria:

   * Adequate tumor tissue from primary tumor resection or biopsy for central pathology review (i.e., B7-H3 expression evaluation by immunohistochemistry [IHC] or H3K27M mutation if pontine lesion)
   * Has a diagnosis of diffuse midline glioma that harbors a mutation associated with this entity (e.g. H3K27M)
   * Has presumptive/suspected brainstem high-grade neoplasm with available imaging for central imaging review
5. Life expectancy of > 12 weeks
6. Adult patient, parent or legal guardian can understand and is willing to sign a written informed consent document according to institutional guidelines

Exclusion Criteria: Screening Eligibility All Participants

1. Participant has other clinically significant medical disorders (e.g. serious infections or significant cardiac, pulmonary, hepatic, psychiatric, or other organ dysfunction) that could compromise their ability to tolerate protocol therapy or would interfere with study procedure.

Inclusion Criteria: Procurement and T-cell Production Eligibility

1. Age ≤ 21 years of age
2. Primary CNS tumor with measurable or evaluable disease and meets criteria for either Cohort A or B:

   * Cohort A: relapsed/refractory non-brainstem CNS primary tumor AND tumor is B7-H3 positive
   * Cohort B: Diffuse midline glioma AND tumor is:

     * B7-H3 positive if non-pontine
     * OR H3K27-altered diffuse midline pontine glioma
     * OR radiographically-confirmed classic/typical DIPG
3. Estimated life expectancy of >12 weeks
4. Karnofsky or Lansky performance score ≥50
5. Participant of childbearing/child-fathering potential agrees to use contraception
6. For females of childbearing age:

   * Not pregnant with negative serum pregnancy test
   * Not lactating with intent to breastfeed
7. Chemotherapy/biologic therapy must be discontinued ≥ 7 days prior to enrollment
8. The last dose of antibody therapy (including check point inhibitor) must be at least 3 half-lives or 30 days, whichever is shorter, from the time of enrollment
9. At least 30 days from most recent cell infusion prior to enrollment.
10. All systemically administered corticosteroid therapy must be stable or decreasing for ≥1 week prior to enrollment, with a maximum dexamethasone dose of 2.8 mg/m^2/day
11. Meets eligibility for apheresis, or has an apheresis product previously collected at a FACT-accredited program
12. Adult patient, parent or legal guardian can understand and is willing to sign a written informed consent document according to institutional guidelines

Exclusion Criteria: Procurement and T-cell Production Eligibility

1. Known primary immunodeficiency or acquired immunodeficiency.
2. Known HIV positivity
3. Severe intercurrent bacterial, viral or fungal infection (e.g. active hepatitis B or C infection or adenovirus infection).
4. Rapidly progressive disease
5. Known underlying medical condition for which participation in this trial would not be in the best interest of the participant or that could prevent, limit or confound protocol assessments.
6. Adult patient, Parent, or legal guardian is unwilling or unable to provide consent for participation in a 15 year long-term follow up study.

Inclusion Criteria: Treatment Eligibility

Cohort A

* Relapsed/refractory non-brainstem CNS primary tumor
* Tumor must be considered B7-H3 positive

Cohort B

* Diffuse Midline Glioma - Must meet one of the following criteria

  * Tumor is considered B7-H3 positive
  * H3K27-altered diffuse midline pontine glioma
  * Radiographically-confirmed classic/typical DIPG
* Must complete standard radiation prior to Loc3CAR treatment and be a minimum of 6 weeks post-completion of radiation therapy

All participants

1. Age ≤ 21 years old
2. Primary CNS tumor with measurable or evaluable disease
3. Available autologous T-cell product that has met GMP release criteria
4. Participant has a CNS reservoir catheter (e.g., Ommaya) or programmable shunt
5. First CAR T cell infusion is planned/scheduled ≥ 5 days from CNS surgery, including catheter placement
6. The following treatments must be discontinued for the specified duration prior to treatment enrollment:

   * Radiation therapy: ≥ 6 weeks
   * Bevacizumab: ≥ 28 days
   * Cytotoxic chemotherapy: ≥ 21 days
   * Biologic agents: ≥ 7 days
   * Antibody therapy: ≥ 3 half-lives or 30 days (whichever is shorter)
   * Cellular therapy: ≥ 30 days
   * Investigational agent: ≥ 3 half-lives or 30 days (whichever is shorter)
   * Corticosteroids: All systemically administered therapy must be stable or decreasing for ≥ 1 week prior to enrollment, with a maximum dexamethasone dose of 2.8 mg/m^2/day. Corticosteroid physiologic replacement therapy for management of pituitary/adrenal axis insufficiency and/or topical administration (e.g. inhaled or dermatologic) is allowed.
7. Estimated life expectancy of >8 weeks
8. Karnofsky or Lansky performance score ≥ 50
9. Echocardiogram with a left ventricular ejection fraction ≥ 50%
10. Adequate renal function defined as calculated creatinine clearance or radioisotope GFR ≥ 50 mL/min/1.73m^2.
11. Adequate pulmonary function defined as forced vital capacity (FVC) ≥50% of predicted value or pulse oximetry ≥90% on room air.
12. Total Bilirubin ≤3 times the upper limit of normal for age.
13. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤5 times the upper limit of normal for age.
14. Hemoglobin >8.0 g/dL (can be transfused).
15. Platelet count >50,000/mm^3 (can be transfused).
16. Absolute neutrophil count (ANC) ≥1000/uL.
17. Taking anti-seizure medication, or agrees to initiate anti-seizure medication prior to starting study therapy.
18. Has recovered from all NCI CTAE grade III-IV, non-hematologic acute toxicities from prior therapy.
19. Male participants of child-fathering potential agree to use contraception
20. Female participants of childbearing potential:

    * Negative serum pregnancy test within 7 days prior to infusion
    * Not lactating with intent to breastfeed
    * If sexually active, agrees to use birth control until 3 months after T-cell infusion. Male partners should use a condom
21. Adult patient, parent or legal guardian can understand and is willing to sign a written informed consent document according to institutional guidelines

Exclusion Criteria: Treatment Eligibility-All Participants

1. Participant has a non-programmable ventricular shunt that could compromise study therapy
2. Participant has a reservoir catheter or shunt in a location that could compromise study therapy or patient safety
3. Known primary immunodeficiency or acquired immunodeficiency.
4. Known HIV positivity
5. Severe intercurrent bacterial, viral or fungal infection
6. Myocardial infarction, unstable angina, New York Heart Association class III and IV congestive heart failure, myocarditis, or ventricular arrhythmias requiring medication within 6 months prior to study entry
7. Receiving therapy as outlined above during the 'wash-out' period
8. Rapidly progressing disease
9. Received any live vaccines within 30 days
10. Known underlying medical condition for which participation in this trial would not be in the best interest of the participant or that could prevent, limit or confound protocol assessments
11. Adult patient, Parent, or legal guardian is unwilling or unable to provide consent for participation in a 15 year long-term follow up study
12. Evidence of uncontrolled hypertension. Anti-hypertensive medications are permitted if on a stable dose.
13. Uncontrolled seizures

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-04-27 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Four (4) weeks after the first B7-H3-CAR T-cell infusion or 7 days after the fourth B7-H3-CAR T cell infusion, whichever is longer
  To determine the maximum tolerated dose for the locoregional delivery of autologous B7-H3-CAR T cells in patients with recurrent/refractory B7-H3- positive primary CNS tumors (Cohort A) or diffuse midline glioma (DMG) (Cohort B).

SECONDARY OUTCOMES:
Radiographic response | Four (4) weeks post B7-H3-CAR T-cell infusion
  To assess the efficacy, defined as sustained objective response, partial response (PR) or complete response (CR), observed anytime on active treatment with B7-H3-CAR T cells in patients with relapsed/refractory B7-H3+ primary CNS tumors (Cohort A) or DMG (Cohort B).

CONTACTS AND LOCATIONS:
Overall Officials: Christopher DeRenzo, MD, Principal Investigator — St. Jude Children's Research Hospital; Kelsey Bertrand, MD, MSc, Principal Investigator — St. Jude Children's Research Hospital; Giedre Krenciute, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols
- See also: St. Jude Brain Tumor Studies — http://www.stjude.org/research/clinical-trials.html#c671955e2f6ffa4a5f9cd8cf39931465e1f28ef99042...